CLINICAL TRIAL: NCT04480268
Title: PAXG Out in the Country
Acronym: OINC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Michele Reni, MD, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PACT31
Record Dates: First submitted 2020-07-14; First posted 2020-07-21 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Combination chemotherapy; PAXG
MeSH Terms: interventions — Cisplatin; 130-nm albumin-bound paclitaxel; Capecitabine; Gemcitabine; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: PAXG regimen (cisplatin, nab-paclitaxel, capecitabine, gemcitabine) chemotherapy — The PAXG regimen includes:
  * nab-paclitaxel 150 mg/m2 on day 1 and 15 of each cycle;
  * cisplatin 30 mg/m2 on day 1 and 15 of each cycle;
  * capecitabine 1250 mg/m2 on 1 day to 28 of each cycle;
  * gemcitabine 800 mg/m2 on day 1 and 15 of each cycle. Each cycle lasts 28 days. Patients are treated until maximal response, disease progression or unacceptable toxicity.

SUMMARY:
The objective of this study is to assess the reproducibility of PAXG regimen as first-line/primary chemotherapy in daily clinical practice in Pancreatic Ductal Adenocarcinoma (PDAC) borderline resectable, locally advanced or metastatic patients out of a large volume center.

DETAILED DESCRIPTION:
Pancreatic Ductal Adenocarcinoma (PDAC) is one of the most lethal malignancies, with a 5-year overall survival (OS) rate for all stages combined lower than 10%, decreasing to 3% in advanced disease. Additionally, PDAC is expected to become the 2nd leading cause for cancer-related death by 2030. Chemotherapy still represents the only therapeutic option in most cases, since 70% of PDAC patients exhibit metastatic or locally advanced disease at diagnosis. Concerning metastatic PDAC patients, combination chemotherapy has resulted in improved survival compared with single-agent treatment. Based on promising phase I/II studies, the PAXG regimen (cisplatin, nab-paclitaxel, capecitabine and gemcitabine) has been recommended for first-line treatment of metastatic PDAC patients in the 2019 edition of Associazione Italiana Oncologia Medica (AIOM) guidelines. Also, this regimen was approved by the Agenzia Italiana del Farmaco (AIFA) as first therapy of borderline-resectable, locally advanced and metastatic PDAC patients with good performance status (ECOG 0-1) and age 18-75 years.

Description of the intervention (schedule of visits):

All PDAC patients who are treated with PAXG regimen as first-line/primary chemotherapy at the participating institutions from January 1st 2020 to December 31st 2020 according to inclusion and exclusion criteria will be included in the present study.

Power size calculation:

The sample size will be as large as possible with a competitive enrollment. All patients treated by the PAXG regimen during 2020 in the participating institutions will be included into the trial. The investigators hypothesize that at least 175 patients (60% metastatic and 40% non-metastatic) from about 30 Italian centers will be enrolled by the end of the year. Such a sample size, or a larger one, will allow to compute in both groups a 95% confident interval of the 1-year OS with at least 10% margin of error, assuming to observe a (target) 1-year OS of 60% for metastatic patients and of 80% for non-metastatic. The trial will be considered successful if the target 1-year OS will fall into the corresponding computed 95% CI.

ELIGIBILITY:
Inclusion Criteria:

* cyto/histological diagnosis of pancreatic adenocarcinoma;
* locally advanced and metastatic disease corresponding to clinical stage III-IV according to TNM 8th Ed. 2017 and borderline resectable disease as anatomically defined according to NCCN Guidelines Version 1.2020 - Pancreatic Adenocarcinoma and biologically defined according to the International consensus on definition and criteria of borderline resectable pancreatic ductal adenocarcinoma 2017 (CA 19.9 > 500 IU/ml);
* ECOG Performance Status ≤1;
* adequate bone marrow function (GB ≥ 3500/mm3, neutrophils ≥1500/mm3, platelets ≥ 100000/mm3, Hb ≥10 g/dl), kidney function (serum creatinine < 1.5 mg/dL) and liver function (ALT and AST < 3 ULN and Serum total bilirubin ≤ 1.5 ULN);
* Patient of child-bearing potential must agree to use two medically acceptable methods of contraception (one for the patient and one for the partner) during the study and for 4 months after the last study treatment intake for women and 6 months for men;
* patients must have received at least 1 cycle (28 days) of the PAXG treatment for the disease within the timeframe starting from January 1 2020 to December 31st 2020 ;
* patient information and signed written informed consent.

Exclusion Criteria:

* previous chemotherapy treatment for recurrent disease;
* concurrent treatment with experimental drugs;
* presence of symptomatic brain metastases;
* heart failure, arrhythmia and/or acute myocardial infarction within 6 months prior to the beginning of PAXG treatment;
* women on pregnancy or lactation;
* history of interstitial lung disease;
* history of connective tissue diseases (systemic lupus erythematosus, systemic sclerosis, etc. ).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival at 1 year (PFS-1yr) | 12 months after the diagnosis
  Primary aim of the study is to evaluate the proportion of patients alive after 1 year from registration

SECONDARY OUTCOMES:
Biochemical Response | 12 months after the diagnosis
  To evaluate the CA19-9 response rate
Radiological Response | 12 months after the diagnosis
  To evaluate the RECIST radiological response
Toxicity profile | 12 months after the diagnosis
  To evaluate drugs toxicity and safety according to according to the "Common Toxicity Criteria" defined by NCI (US) and integrated by NCIC (Canada) version 5.0
Progression-free survival (PFS) | 5 year after the diagnosis
  To evaluate the progression-free survival (PFS), defined as the time between the date of registration and the date of documented radiological PD or death from any cause, whichever occurs first, or the date of last follow-up or last available tumour assessment if no further follow-up for disease progression is performed.
Overall Survival (OS) | 5 year after the diagnosis
  To evaluate the overall survival (OS), defined as time between the date of registration and the date of death for any cause or the date they were last known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Reni, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (30):
- Italy (30):
  - IRCCS Centro di Riferimento Oncologico (CRO), Aviano
  - Istituto dei tumori Giovanni Paolo II, Bari
  - AULSS 1 di Belluno, Belluno
  - ASST Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera Policlinico Sant'Orsola-Malpighi, Bologna
  - Azienda Ospedaliera AOU di Cagliari, Cagliari
  - Ospedale di Carpi, Carpi
  - USL Toscana Nord Ovest, Carrara
  - Fondazione Istituto Giglio, Cefalù
  - Ospedaliera Sant' Anna di Como Asst Lariana, Como
  - Azienda Ospedaliera Universitaria Ospedali Riuniti di Foggia, Foggia
  - ASST Rhodense, Garbagnate
  - Ospedale Moriggia Pelascini, Gravedona
  - Ospedale Generale Provinciale di Macerata, Macerata
  - Irccs Irst, Meldola
  - ASST Melegnano e Della Martesana, Melegnano
  - IRCCS San Raffaele Medical Oncology Unit, Milan
  - Istituto Oncologico Veneto IRCCS, Padua
  - Ospedale Civico di Palermo, Palermo
  - Azienda Ospedaliera di Parma, Parma
  - Azienda Ospedaliera di Piacenza, Piacenza
  - Giovanni Paolo II-Maria Paternò, Ragusa
  - Azienda Ospedaliera Universitaria San Giovanni di Dio e Ruggi D'Aragona, Salerno
  - AULSS 4 Veneto Orientale, San Donà di Piave
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Azienda Ospedaliera Ordine Mauriziano, Torino
  - Presidio Ospedaliero Molinette, Torino
  - Azienda Sanitaria Universitaria Integrata, Udine
  - ASST Sette Laghi, Varese
  - Ospedale San Bortolo Azienda ULSS8 Berica-Distretto Est, Vicenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reni M, Cereda S, Rognone A, Belli C, Ghidini M, Longoni S, Fugazza C, Rezzonico S, Passoni P, Slim N, Balzano G, Nicoletti R, Cappio S, Doglioni C, Villa E. A randomized phase II trial of two different 4-drug combinations in advanced pancreatic adenocarcinoma: cisplatin, capecitabine, gemcitabine plus either epirubicin or docetaxel (PEXG or PDXG regimen). Cancer Chemother Pharmacol. 2012 Jan;69(1):115-23. doi: 10.1007/s00280-011-1680-2. Epub 2011 May 28. PMID 21626049
- [Background] Reni M, Balzano G, Zanon S, Passoni P, Nicoletti R, Arcidiacono PG, Pepe G, Doglioni C, Fugazza C, Ceraulo D, Falconi M, Gianni L. Phase 1B trial of Nab-paclitaxel plus gemcitabine, capecitabine, and cisplatin (PAXG regimen) in patients with unresectable or borderline resectable pancreatic adenocarcinoma. Br J Cancer. 2016 Jul 26;115(3):290-6. doi: 10.1038/bjc.2016.209. Epub 2016 Jul 12. PMID 27404453
- [Background] Reni M, Zanon S, Peretti U, Chiaravalli M, Barone D, Pircher C, Balzano G, Macchini M, Romi S, Gritti E, Mazza E, Nicoletti R, Doglioni C, Falconi M, Gianni L. Nab-paclitaxel plus gemcitabine with or without capecitabine and cisplatin in metastatic pancreatic adenocarcinoma (PACT-19): a randomised phase 2 trial. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):691-697. doi: 10.1016/S2468-1253(18)30196-1. Epub 2018 Jul 7. PMID 30220407
- [Background] Reni M, Zanon S, Balzano G, Passoni P, Pircher C, Chiaravalli M, Fugazza C, Ceraulo D, Nicoletti R, Arcidiacono PG, Macchini M, Peretti U, Castoldi R, Doglioni C, Falconi M, Partelli S, Gianni L. A randomised phase 2 trial of nab-paclitaxel plus gemcitabine with or without capecitabine and cisplatin in locally advanced or borderline resectable pancreatic adenocarcinoma. Eur J Cancer. 2018 Oct;102:95-102. doi: 10.1016/j.ejca.2018.07.007. Epub 2018 Aug 24. PMID 30149366